CLINICAL TRIAL: NCT02722954
Title: A Phase 1b, Open-Label, Dose Escalation and Expansion Study of Demcizumab Plus Pembrolizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1b Study of Demcizumab Plus Pembrolizumab in Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M18-008
Record Dates: First submitted 2016-03-07; First posted 2016-03-30 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
Keywords: malignancy; metastatic; Demcizumab; Pembrolizumab; Phase 1b
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — demcizumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Demcizumab and Pembrolizumab (Experimental): Demcizumab will be administered prior to pembrolizumab
  Interventions: Drug: Demcizumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Demcizumab — Drug: Demcizumab at starting dose of 2.5mg/kg administered intravenously (IV).
  Other Names: OMP-21M18
Drug: Pembrolizumab — Drug: Pembrolizumab administered 2mg/kg IV every 3 weeks

SUMMARY:
The purpose of this study is to test the efficacy and safety of an experimental drug, demcizumab, when given in combination with pembrolizumab. Demcizumab is a humanized monoclonal antibody and was developed to target cancer stem cells. Demcizumab may block the growth of cancer stem cells, the remaining cancer cells, and it may also impair the productive growth of new blood vessels, which tumors need to grow and spread.

This study is sponsored by OncoMed Pharmaceuticals, which is referred to as OncoMed or the Sponsor in this consent form.

DETAILED DESCRIPTION:
This is an open-label, Phase 1b dose escalation and expansion study of demcizumab plus pembrolizumab designed to evaluate the safety, efficacy and pharmacokinetics of demcizumab in combination with pembrolizumab in patients with advanced or metastatic solid tumors. This study consists of a screening period, a treatment period and a post-treatment follow up period in which patients will be followed for survival for approximately 12 months. Patients will be enrolled in two stages: a dose-escalation stage and an expansion phase.

Approximately 42 patients will be enrolled in this study at approximately 10 study centers in the United States (U.S) and Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Measurable disease per response evaluation criteria in solid tumors (RECIST) v1.1
2. Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue, either fresh core-needle-biopsied or archived
3. Age >21 years
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Adequate organ and marrow function
6. For women of childbearing potential and men with partners of childbearing potential, agreement (by patient and/or partner) to use two effective forms of contraception from study entry through at least 6 months after the termination visit.
7. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Treatment with any anti-cancer therapy, including radiotherapy, chemotherapy, biologic therapy, or herbal therapy within 3 weeks or 5 half-lives (for systemic agents) whichever is shorter
2. Receiving any other investigational agents or any other anti-cancer therapy
3. Active infections requiring antibiotics
4. Patients with brain metastases (treated or untreated) leptomeningeal disease, uncontrolled seizure disorder, or active neurologic disease
5. History of interstitial lung disease or active, non-infectious pneumonitis that required oral or intravenous corticosteroids
6. Prior radiation to the chest wall or mediastinum if the radiation field involves the heart
7. Significant intercurrent illness that will limit the patient's ability to participate in the study or may result in their death over the next 18 months
8. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment, or anticipation of need for major surgical procedure during the course of the study
9. Pregnant or nursing women
10. New York Heart Association Classification II, III, or IV
11. Acute prior study treatment related toxicity (except alopecia) that has not resolved to Grade < or = to 1 unless it has been deemed stable by the investigator
12. Inability to comply with study and follow up procedure

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) of demcizumab given in combination with pembrolizumab | Subjects will be treated and observed for DLT through the end of the first cycle (Days 1-22)
  The maximum tolerated dose (MTD) or maximum administered dose (MAD) will be determined in patients treated with demcizumab in combination with pembrolizumab

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of demcizumab and pembrolizumab | Plasma sample for Pharmacokinetics (PK) analysis to be obtained on Days 1, 22, 43 then at every other cycle (each cycle is 21 days) until 12 weeks post treatment termination, an average of 1 year
  peak plasma concentration

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - University of Michigan Health System, Ann Arbor, Michigan
  - Columbia University Medical Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The START Center for Cancer Care, San Antonio, Texas
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom